CLINICAL TRIAL: NCT03520569
Title: Effect of Hyperglycemia on Microvascular Perfusion in Healthy Adults
Acronym: EJB050
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Eugene Barrett, Prinicipal Investigator, University of Virginia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 19948; T32DK007646 (NIH)
Record Dates: First submitted 2018-03-08; First posted 2018-05-09 (Actual); Results first posted 2022-05-13 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2022-04

CONDITIONS: Vascular Stiffness; Insulin Sensitivity
MeSH Terms: conditions — Insulin Resistance | interventions — Octreotide; Insulin; Glucose; Solutions

STUDY DESIGN:
Intervention Model Description: Each subject is studied 4 times in a randomized sequential order
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Octreotide- Euglycemia (Active Comparator): octreotide is 30 ng/kg/min x 240 min insulin 0.15mU/kg/min x 240 min Dextrose 20% at variable rate to maintain euglycemia for 240 min
  Interventions: Drug: Octreotide; Drug: Insulin; Drug: Dextrose 20% solution
- Octreotide - Euglycemia- insulin clamp (Active Comparator): octreotide is 30 ng/kg/min x 330 min insulin 0.15mU/kg/min x 210 min insulin 1.0mU/kg/min x 120 min Dextrose 20% at variable rate to maintain euglycemia for 330 min
  Interventions: Drug: Octreotide; Drug: Insulin; Drug: Dextrose 20% solution
- Octreotide- hyperglycemia (Active Comparator): octreotide is 30 ng/kg/min x 330 min insulin 0.15mU/kg/min x 330 min Dextrose 20% at variable rate to maintain euglycemia for 90 min Dextrose 20% at variable rate to maintain hyperglycemia for 240 min
  Interventions: Drug: Octreotide; Drug: Insulin; Drug: Dextrose 20% solution
- Octreotide- hyperglycemia - insulin clamp (Active Comparator): octreotide is 30 ng/kg/min x 330 min insulin 0.15mU/kg/min x 210 min insulin 1.0mU/kg/min x 120 min Dextrose 20% at variable rate to maintain euglycemia for 90 min Dextrose 20% at variable rate to maintain hyperglycemia for 240 min
  Interventions: Drug: Octreotide; Drug: Insulin; Drug: Dextrose 20% solution

INTERVENTIONS:
Drug: Octreotide — we are using it to block insulin secretion from the pancreas
Drug: Insulin — we are using to replace basal insulin and in two protocols to raise insulin concentrations during the insulin clamp
Drug: Dextrose 20% solution — We are using dextrose to maintain glycemia level

SUMMARY:
The investigators are studying the effects of Hyperglycemia on vascular function and insulin sensitivity on healthy adults

DETAILED DESCRIPTION:
The investigators will study 22 healthy subjects (18-35 yrs) four times as follows:

1. Saline + Octreotide + euglycemia;
2. Octreotide + hyperglycemia;
3. Octreotide + hyperglycemia + insulin clamp and
4. Octreotide + Euglycemia + insulin clamp.

The sequence of admissions will be assigned randomly. The investigators will assess function in conduit (pulse wave velocity-PWV, augmentation index-AI and flow-mediated dilation-FMD), resistance (post-ischemic flow velocity-PIFV) and heart and skeletal muscle microvascular (contrast enhanced ultrasound-CEU) vessels.

This work will:

a) identify whether vascular stiffness and indices of NO action are impaired throughout the arterial tree with hyperglycemia.

ELIGIBILITY:
Inclusion Criteria:

* Healthy with no chronic illness
* Age 18-35
* Normal BMI (18-25)
* Normal screening labs or no clinically significant values

Exclusion Criteria:

* First degree relative with Type 2 Diabetes
* Smoking presently or in the past 6 months
* Medications that affect the vasculature
* Overweight or other indications of insulin resistance
* Elevated LDL cholesterol > 160
* Elevated BP > 140/90
* History of congestive heart failure, ischemic heart disease, severe pulmonary disease, liver or kidney disease, bleeding disorders
* Any vascular disease such as myocardial infarction, stroke, peripheral vascular disease
* Presence of an intracardiac or intrapulmonary shunt (we will screen for this by auscultation during the physical exam by PI).
* Pregnant or breastfeeding.
* Known hypersensitivity to perflutren (contained in Definity)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2019-02-04 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Deedwania P, Kosiborod M, Barrett E, Ceriello A, Isley W, Mazzone T, Raskin P. Hyperglycemia and acute coronary syndrome: a scientific statement from the American Heart Association Diabetes Committee of the Council on Nutrition, Physical Activity, and Metabolism. Anesthesiology. 2008 Jul;109(1):14-24. doi: 10.1097/ALN.0b013e31817dced3. PMID 18580168
- [Background] Brownlee M. Biochemistry and molecular cell biology of diabetic complications. Nature. 2001 Dec 13;414(6865):813-20. doi: 10.1038/414813a. PMID 11742414
- [Background] Giacco F, Brownlee M. Oxidative stress and diabetic complications. Circ Res. 2010 Oct 29;107(9):1058-70. doi: 10.1161/CIRCRESAHA.110.223545. PMID 21030723
- [Background] Brouwers O, Niessen PM, Haenen G, Miyata T, Brownlee M, Stehouwer CD, De Mey JG, Schalkwijk CG. Hyperglycaemia-induced impairment of endothelium-dependent vasorelaxation in rat mesenteric arteries is mediated by intracellular methylglyoxal levels in a pathway dependent on oxidative stress. Diabetologia. 2010 May;53(5):989-1000. doi: 10.1007/s00125-010-1677-0. Epub 2010 Feb 26. PMID 20186387
- [Background] Ceriello A, Taboga C, Tonutti L, Quagliaro L, Piconi L, Bais B, Da Ros R, Motz E. Evidence for an independent and cumulative effect of postprandial hypertriglyceridemia and hyperglycemia on endothelial dysfunction and oxidative stress generation: effects of short- and long-term simvastatin treatment. Circulation. 2002 Sep 3;106(10):1211-8. doi: 10.1161/01.cir.0000027569.76671.a8. PMID 12208795
- [Background] Suzuki K, Watanabe K, Futami-Suda S, Yano H, Motoyama M, Matsumura N, Igari Y, Suzuki T, Nakano H, Oba K. The effects of postprandial glucose and insulin levels on postprandial endothelial function in subjects with normal glucose tolerance. Cardiovasc Diabetol. 2012 Aug 14;11:98. doi: 10.1186/1475-2840-11-98. PMID 22891922
- [Background] Ceriello A, Novials A, Ortega E, Canivell S, La Sala L, Pujadas G, Esposito K, Giugliano D, Genovese S. Glucagon-like peptide 1 reduces endothelial dysfunction, inflammation, and oxidative stress induced by both hyperglycemia and hypoglycemia in type 1 diabetes. Diabetes Care. 2013 Aug;36(8):2346-50. doi: 10.2337/dc12-2469. Epub 2013 Apr 5. PMID 23564922
- [Background] Perkins JM, Joy NG, Tate DB, Davis SN. Acute effects of hyperinsulinemia and hyperglycemia on vascular inflammatory biomarkers and endothelial function in overweight and obese humans. Am J Physiol Endocrinol Metab. 2015 Jul 15;309(2):E168-76. doi: 10.1152/ajpendo.00064.2015. Epub 2015 May 26. PMID 26015434
- [Background] Giugliano D, Marfella R, Coppola L, Verrazzo G, Acampora R, Giunta R, Nappo F, Lucarelli C, D'Onofrio F. Vascular effects of acute hyperglycemia in humans are reversed by L-arginine. Evidence for reduced availability of nitric oxide during hyperglycemia. Circulation. 1997 Apr 1;95(7):1783-90. doi: 10.1161/01.cir.95.7.1783. PMID 9107164
- [Background] Cuypers MH, Kasanardjo JS, Polak BC. Retinal blood flow changes in diabetic retinopathy measured with the Heidelberg scanning laser Doppler flowmeter. Graefes Arch Clin Exp Ophthalmol. 2000 Dec;238(12):935-41. doi: 10.1007/s004170000207. PMID 11196354
- [Background] Horova E, Mazoch J, Hiigertova J, Kvasnicka J, Skrha J, Soupal J, Prazny M. Acute hyperglycemia does not impair microvascular reactivity and endothelial function during hyperinsulinemic isoglycemic and hyperglycemic clamp in type 1 diabetic patients. Exp Diabetes Res. 2012;2012:851487. doi: 10.1155/2012/851487. Epub 2012 Jan 4. PMID 22262970
- [Background] Burgansky-Eliash Z, Barak A, Barash H, Nelson DA, Pupko O, Lowenstein A, Grinvald A, Rubinstein A. Increased retinal blood flow velocity in patients with early diabetes mellitus. Retina. 2012 Jan;32(1):112-9. doi: 10.1097/IAE.0b013e31821ba2c4. PMID 21878846
- [Background] Rattigan S, Clark MG, Barrett EJ. Hemodynamic actions of insulin in rat skeletal muscle: evidence for capillary recruitment. Diabetes. 1997 Sep;46(9):1381-8. doi: 10.2337/diab.46.9.1381. PMID 9287035
- [Background] Chai W, Zhang X, Barrett EJ, Liu Z. Glucagon-like peptide 1 recruits muscle microvasculature and improves insulin's metabolic action in the presence of insulin resistance. Diabetes. 2014 Aug;63(8):2788-99. doi: 10.2337/db13-1597. Epub 2014 Mar 21. PMID 24658303
- [Background] Vincent MA, Dawson D, Clark AD, Lindner JR, Rattigan S, Clark MG, Barrett EJ. Skeletal muscle microvascular recruitment by physiological hyperinsulinemia precedes increases in total blood flow. Diabetes. 2002 Jan;51(1):42-8. doi: 10.2337/diabetes.51.1.42. PMID 11756321
- [Background] Clerk LH, Vincent MA, Jahn LA, Liu Z, Lindner JR, Barrett EJ. Obesity blunts insulin-mediated microvascular recruitment in human forearm muscle. Diabetes. 2006 May;55(5):1436-42. doi: 10.2337/db05-1373. PMID 16644702
- [Background] Clerk LH, Vincent MA, Barrett EJ, Lankford MF, Lindner JR. Skeletal muscle capillary responses to insulin are abnormal in late-stage diabetes and are restored by angiotensin-converting enzyme inhibition. Am J Physiol Endocrinol Metab. 2007 Dec;293(6):E1804-9. doi: 10.1152/ajpendo.00498.2007. Epub 2007 Oct 2. PMID 17911341
- [Background] Jahn LA, Hartline L, Rao N, Logan B, Kim JJ, Aylor K, Gan LM, Westergren HU, Barrett EJ. Insulin Enhances Endothelial Function Throughout the Arterial Tree in Healthy But Not Metabolic Syndrome Subjects. J Clin Endocrinol Metab. 2016 Mar;101(3):1198-206. doi: 10.1210/jc.2015-3293. Epub 2016 Jan 12. PMID 26756115
- [Background] Inyard AC, Chong DG, Klibanov AL, Barrett EJ. Muscle contraction, but not insulin, increases microvascular blood volume in the presence of free fatty acid-induced insulin resistance. Diabetes. 2009 Nov;58(11):2457-63. doi: 10.2337/db08-1077. Epub 2009 Aug 12. PMID 19675134
- [Background] Liu J, Jahn LA, Fowler DE, Barrett EJ, Cao W, Liu Z. Free fatty acids induce insulin resistance in both cardiac and skeletal muscle microvasculature in humans. J Clin Endocrinol Metab. 2011 Feb;96(2):438-46. doi: 10.1210/jc.2010-1174. Epub 2010 Nov 3. PMID 21047922
- [Background] Marfella R, Nappo F, De Angelis L, Siniscalchi M, Rossi F, Giugliano D. The effect of acute hyperglycaemia on QTc duration in healthy man. Diabetologia. 2000 May;43(5):571-5. doi: 10.1007/s001250051345. PMID 10855531
- [Background] Glaser N, Ngo C, Anderson S, Yuen N, Trifu A, O'Donnell M. Effects of hyperglycemia and effects of ketosis on cerebral perfusion, cerebral water distribution, and cerebral metabolism. Diabetes. 2012 Jul;61(7):1831-7. doi: 10.2337/db11-1286. Epub 2012 Apr 12. PMID 22498698
- [Background] Wei K, Jayaweera AR, Firoozan S, Linka A, Skyba DM, Kaul S. Quantification of myocardial blood flow with ultrasound-induced destruction of microbubbles administered as a constant venous infusion. Circulation. 1998 Feb 10;97(5):473-83. doi: 10.1161/01.cir.97.5.473. PMID 9490243
- [Background] Chai W, Liu J, Jahn LA, Fowler DE, Barrett EJ, Liu Z. Salsalate attenuates free fatty acid-induced microvascular and metabolic insulin resistance in humans. Diabetes Care. 2011 Jul;34(7):1634-8. doi: 10.2337/dc10-2345. Epub 2011 May 26. PMID 21617098
- [Background] Scognamiglio R, Negut C, De Kreutzenberg SV, Tiengo A, Avogaro A. Postprandial myocardial perfusion in healthy subjects and in type 2 diabetic patients. Circulation. 2005 Jul 12;112(2):179-84. doi: 10.1161/CIRCULATIONAHA.104.495127. Epub 2005 Jul 5. PMID 15998667
- [Background] Abdelmoneim SS, Hagen ME, Mendrick E, Pattan V, Wong B, Norby B, Roberson T, Szydel T, Basu R, Basu A, Mulvagh SL. Acute hyperglycemia reduces myocardial blood flow reserve and the magnitude of reduction is associated with insulin resistance: a study in nondiabetic humans using contrast echocardiography. Heart Vessels. 2013 Nov;28(6):757-68. doi: 10.1007/s00380-012-0305-y. Epub 2012 Nov 23. PMID 23180239
- [Background] Eggleston EM, Jahn LA, Barrett EJ. Hyperinsulinemia rapidly increases human muscle microvascular perfusion but fails to increase muscle insulin clearance: evidence that a saturable process mediates muscle insulin uptake. Diabetes. 2007 Dec;56(12):2958-63. doi: 10.2337/db07-0670. Epub 2007 Aug 24. PMID 17720897
- [Background] DeFronzo RA, Tobin JD, Andres R. Glucose clamp technique: a method for quantifying insulin secretion and resistance. Am J Physiol. 1979 Sep;237(3):E214-23. doi: 10.1152/ajpendo.1979.237.3.E214. PMID 382871
- [Background] Cardillo C, Nambi SS, Kilcoyne CM, Choucair WK, Katz A, Quon MJ, Panza JA. Insulin stimulates both endothelin and nitric oxide activity in the human forearm. Circulation. 1999 Aug 24;100(8):820-5. doi: 10.1161/01.cir.100.8.820. PMID 10458717
- [Derived] Horton WB, Jahn LA, Hartline LM, Aylor KW, Patrie JT, Barrett EJ. Insulin increases central aortic stiffness in response to hyperglycemia in healthy humans: A randomized four-arm study. Diab Vasc Dis Res. 2021 Mar-Apr;18(2):14791641211011009. doi: 10.1177/14791641211011009. PMID 33908285
- [Derived] Horton WB, Jahn LA, Hartline LM, Aylor KW, Patrie JT, Barrett EJ. Acute hyperglycaemia enhances both vascular endothelial function and cardiac and skeletal muscle microvascular function in healthy humans. J Physiol. 2022 Feb;600(4):949-962. doi: 10.1113/JP281286. Epub 2021 Feb 2. PMID 33481251

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 20 potential study participants were screened for eligibility
Pre-assignment Details: 15 participants were ultimately enrolled. Five potential subjects failed to meet inclusion criteria and were subsequently excluded from the study.
Groups:
- All Participants: All participants enrolled who completed at least one arm of the crossover assignment.
Period: Overall Study
Arm/Group | All Participants
Started | 15
Octreotide-Euglycemia | 13
Octreotide-Euglycemia-Insulin Clamp | 14
Octreotide-Hyperglycemia | 10
Octreotide-Hyperglycemia-Insulin Clamp | 12
Completed | 14
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: 15 subjects participated in the study - 1 person withdrew
Groups:
- All Participants: all participants who completed the study
Arm/Group | All Participants
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 24 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  caucasian | 13
  african american | 1
  asian | 1
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Change in Flow Mediated Dilation (FMD) Between Baseline and After 2 Hour Insulin Clamp
Description: Flow mediated dilation measures the change in brachial diameter in response to 5 minutes of ischemia using B-mode ultrasound. It provides an index of nitric oxide generation by the endothelium .
Time Frame: baseline and after 2 hour insulin clamp
Measure: Mean (Standard Deviation); unit: % change
Arm/Group | Octreotide- Euglycemia | Octreotide - Euglycemia- Insulin Clamp | Octreotide- Hyperglycemia | Octreotide- Hyperglycemia - Insulin Clamp
Number analyzed (Participants) | 13 | 14 | 10 | 12
% change | 11.8 (4.4) | 11.8 (4) | 8.9 (4.3) | 8.95 (4.5)

2. Secondary Outcome: Change in Augmentation Index Between Baseline and After 2 Hour Insulin Clamp
Description: The augmentation index (AIx) measured at the radial artery is a measure of systemic arterial stiffness, and is defined as the ratio of augmentation (Δ P) to central pulse pressure and expressed as percent. AIx = (ΔP/PP) x 100, where P = pressure and PP = Pulse Pressure. Higher percentages indicate increased arterial stiffness.
Time Frame: baseline and after 2 hour insulin clamp
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Octreotide- Euglycemia | Octreotide - Euglycemia- Insulin Clamp | Octreotide- Hyperglycemia | Octreotide- Hyperglycemia - Insulin Clamp
Number analyzed (Participants) | 13 | 14 | 10 | 12
percentage | -4.15 (11.72) | -2.23 (12.33) | -4.80 (12.13) | -8.45 (9.16)

3. Secondary Outcome: Change in Pulse Wave Velocity (PWV) Between Baseline and After 2 Hour Insulin Clamp
Description: The time required for a blood pressure wave to travel from the carotid to the femoral artery was measured in meter/sec. This is a measurement of central artery stiffness. Higher numbers indicate stiffer vessels
Time Frame: baseline and after 2 hour insulin clamp
Measure: Mean (Standard Deviation); unit: m/sec
Arm/Group | Octreotide- Euglycemia | Octreotide - Euglycemia- Insulin Clamp | Octreotide- Hyperglycemia | Octreotide- Hyperglycemia - Insulin Clamp
Number analyzed (Participants) | 13 | 14 | 10 | 12
m/sec | 5.21 (0.64) | 5.06 (0.76) | 4.79 (0.79) | 5.07 (0.67)

ADVERSE EVENTS:
Time Frame: 20 months
Arm/Group | Octreotide- Euglycemia | Octreotide - Euglycemia- Insulin Clamp | Octreotide- Hyperglycemia | Octreotide- Hyperglycemia - Insulin Clamp
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/14 | 0/10 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/14 | 0/10 | 0/12
Other Adverse Events (participants affected / at risk) | 0/13 | 0/14 | 0/10 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-16): https://cdn.clinicaltrials.gov/large-docs/69/NCT03520569/Prot_SAP_000.pdf